CLINICAL TRIAL: NCT06255860
Title: SARS-COV-2 (virus Responsible of COVID-19) Reinfection and Multisystem Inflammatory Syndrome in Children (MIS-C) Risk: Matched Case-control Study
Brief Title: COVID-19 and Multisystem Inflammatory Syndrome in Children (MIS-C) Risk / World Health Organization (WHO)
Acronym: REPI
Status: Completed | Type: Observational
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Sponsor
Other Study IDs: REPI
Record Dates: First submitted 2024-02-07; First posted 2024-02-13 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Sars-CoV-2 Infection; MIS-C
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- children with MIS-C: hospitalized children with MIS-C
- SARS-CoV-2 infection: non hospitalized children infected with SARS-CoV-2 treated by outpatient care

SUMMARY:
This study is a multicenter, international, non interventional, retrospective study about SARS-CoV-2 and Multisystem Inflammatory Syndrome (MIS-C) reinfection risk in children.

DETAILED DESCRIPTION:
This study is based to data collection of cases (patients with MIS-C) compare to controls (patients with SARS-CoV-2 infection) occurring between 01 sep 2021 and 30 apr 2022. For this study cases and controls group will be matched for analyses.

The main of this study is to evaluate the difference of risk of occurrence of MIS-C between a first SARS-CoV-2 infection and a reinfection with SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

group 1: cases

* Patients with MIS-C (following SARS CoV-2 infection)
* Hospitalised between the 01 sep 2021 and 30 apr 2022
* Under 18 years of age
* Not vaccinated for SARS-CoV-2

group 2: controls

* Patients not hospitalised, treated by outpatient care
* With documented SARS-CoV-2 infection between the 01 sep 2021 and 30 apr 2022
* Matched with a case on age (+/- 6 months), gender and country
* Not vaccinated for SARS-CoV-2

Exclusion Criteria:

- Refusal to participate by patient relative or legal representative

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children with SARS-CoV-2 and children with MIS-C between the 01 sep 2021 and 30 apr 2022 period
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
proportion of MIS-C cases occurred after first SARS-CoV-2 infection | 8 months
  Assessment of risk of MIS-C after first SARS-CoV-2 infection
proportion of MIS-C cases occurred after SARS-CoV-2 reinfection | 8 months
  Assessment of risk of MIS-C after SARS-CoV-2 reinfection
Proportion of SARS-CoV-2 reinfection after first SARS-CoV-2 infection | 8 months
  Assessment of risk of SARS-CoV-2 reinfection after first SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Levy, Physician, Study Director — Association Clinique Thérapeutique Infantile du val de Marne; Naim Ouldali, Physician, Principal Investigator — Hôpital Robert Debré AP-HP, Paris 19
Locations (1):
- ACTIV, Créteil, France

IPD SHARING:
Plan to Share IPD: No